CLINICAL TRIAL: NCT01994954
Title: A Randomized Trial of Outpatient Oxygen Weaning Strategies in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Bay State Medical Center (Unknown); UConn Health (Other); University of Vermont Medical Center (Other); Connecticut Children's Medical Center (Other); Patient-Centered Outcomes Research Institute (Other); University of Kentucky (Other); Boston Children's Hospital (Other); Dartmouth-Hitchcock Medical Center (Other); Tufts Medical Center (Other); Westchester Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IP00009772
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Premature Infants
Keywords: newborn intensive care unit; NICU; supplemental oxygen
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A:Standard therapy (No Intervention): Infants' oxygen will be increased, decreased, or maintained based on brief structured assessments during monthly clinic visits. Polysomnograms will be utilized prior to final discontinuation of oxygen. RHO will only be utilized on the night prior to and during the polysomnogram to compare these two modalities.
- Arm B:RHO (Experimental): Infants will have the same monthly clinic assessments as in Arm A, but also will utilize RHO to potentially increase, decrease or maintain oxygen between monthly visits.
  Parents will transmit a minimum of 4 days of stored RHO data (min 8 hrs per day) every 4-7 days. Changes in oxygen needs will be made based on standardized objective criteria. To determine discontinuation of oxygen, RHO will be utilized instead of polysomnography.
  Interventions: Other: RHO

INTERVENTIONS:
Other: RHO — Recorded oximetry data will be downloaded from home oximeters, analyzed, and used to assist in supplemental oxygen weaning decisions.
  Arms: Arm B:RHO

SUMMARY:
The investigators hypothesize that Recorded Home Oximetry (RHO) utilization will not increase rates of respiratory-related re-hospitalizations and ED visits, and will not impair growth compared to standard oxygen management protocols.

Evidence-based specific consensus guidelines for home regulated oxygen management do not currently exist. Current strategies for infants requiring outpatient supplemental home oxygen include brief checks of oxygen status during monthly clinic visits. Although the infants stay on monitors, no data in between visits is obtained to ensure that infants can maintain oxygen levels after weans are made. Before finally allowing oxygen to be removed, many centers also require an overnight sleep study in the hospital, to make sure that the infant's oxygen levels stay safe when the infant is in deep sleep. Because these methods rely solely on assumptions rather than individually recorded data, an infant's time on supplemental oxygen may be prolonged or insufficient. This study will evaluate both the currently used accepted therapy and a method of weaning that involves recording and sending oxygen data for analysis in between clinic visits.

Premature infants who require home oxygen therapy at time of discharge who meet eligibility criteria will be randomized into two arms:

Arm A ("Standard therapy"): Infants' oxygen will be increased, decreased, or maintained based on brief structured assessments during monthly clinic visits.

Arm B (Recorded Home Oximetry (RHO)): Infants will have the same monthly clinic assessments as in Arm A, but also will utilize Recorded Home Oximetry (RHO) to potentially increase, decrease or maintain oxygen between monthly visits.

Parents of all infants will be interviewed using structured quality-of-life questionnaires at the beginning and ending of the oxygen management process. Health care utilization (emergency department visits and rehospitalizations) and growth will be assessed 6 months after discontinuation of oxygen.

The investigators overall objective is to determine whether Recorded Home Oximetry (RHO) can improve caregiver quality of life, and can shorten Home Oxygen Therapy (HOT) duration and eliminate need for polysomnogram, without compromising safety. The investigators will determine respiratory-related re-hospitalizations, emergency department (ED) visits, and growth parameters to confirm safety of the proposed weaning strategies.

ELIGIBILITY:
Inclusion Criteria:

* Infant with birth gestational age ≤ 37 (37 0/7) wks postmenstrual age (PMA) who has requirement for supplemental O2 at time of NICU discharge, as determined by primary NICU team.
* Infant receiving pediatric pulmonology care at the Center for Healthy Infant Lung Development
* Parent aged 18 years or older
* English or Spanish-speaking.

Exclusion Criteria:

* Parents whose infants has presence of pulmonary hypertension at enrollment
* Parents whose infant with syndrome or other diagnosis with known high risk for persistent hypoxia (cardiac disease, Trisomy 21, Pierre-Robin Sequence, etc.)
* Parents whose infant has requirement for O2 flow rate > 1 L/min or tracheostomy
* Any infants who also require caffeine at discharge from the NICU

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Rhein, MD, MPH, Principal Investigator — University of Massachusetts, Worcester; Heather White, BS, Study Director — University of Massachusetts, Worcester
Locations (8):
- United States (8):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Kentucky Children's Hospital at University of Kentucky, Lexington, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Boston Children's Hospital Physicians, Valhalla, New York
  - University of Vermont Medical Center, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were screened from November 2013 to December 2017. Subjects were screened either before NICU discharge with anticipation of HOT therapy or at their first pulmonary clinic visit. Each subject was consented at their first outpatient pulmonary clinic or NICU follow-up clinic with a pulmonary component.
Groups:
- Arm B:RHO: Infants will have the same monthly clinic assessments as in Arm A, but also will utilize RHO to potentially increase, decrease or maintain oxygen between monthly visits.
  Parents will transmit a minimum of 4 days of stored RHO data (min 8 hrs per day) every 4-7 days. Changes in oxygen needs will be made based on standardized objective criteria. To determine discontinuation of oxygen, RHO will be utilized instead of polysomnography.
  RHO: Recorded oximetry data will be downloaded from home oximeters, analyzed, and used to assist in supplemental oxygen weaning decisions.
Period: Overall Study
Arm/Group | Arm A:Standard Therapy | Arm B:RHO
Started | 99 | 97
Completed | 74 | 67
Not Completed | 25 | 30
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 9 | 14
Not completed — Physician Decision | 2 | 2
Not completed — Lost to Follow-up | 8 | 10
Not completed — 6 Month Follow-up Not Complete | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A:Standard Therapy | Arm B:RHO | Total
Number analyzed (Participants) | 99 | 97 | 196
Age, Customized [Count of Participants; unit: Participants]
  Less than 1 Year of Age | 99 | 97 | 196
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 33 | 74
  Male | 58 | 64 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 18
  Not Hispanic or Latino | 61 | 65 | 126
  Unknown or Not Reported | 26 | 26 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 13 | 25
  White | 57 | 59 | 116
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 22 | 15 | 37
Region of Enrollment [Number; unit: participants]
  United States | 99 | 97 | 196
Respiratory Support at 36 Weeks [Count of Participants; unit: Participants]
  Mechanical Ventilation | 3 | 6 | 9
  Non-Invasive Positive Pressure (CPAP/HFNC) | 52 | 48 | 100
  Low-Flow Nasal Cannula (LFNC) | 36 | 32 | 68
  Room Air | 2 | 5 | 7
  Unknown | 6 | 6 | 12
Diuretics [Count of Participants; unit: Participants]
  Yes | 52 | 51 | 103
  No | 41 | 38 | 79
  Unknowns | 6 | 8 | 14
Birth Weight [Mean (Standard Deviation); unit: grams] | 938.2 (439.1) | 929.5 (442.6) | 933.9 (439.6)
Gestational Age (wks) [Mean (Standard Deviation); unit: Birth Gestational Age (Weeks)] | 26.9 (2.6) | 26.9 (2.7) | 26.9 (2.6)
Length of NICU Stay (days) [Mean (Standard Deviation); unit: days] | 97.7 (33.4) | 104.4 (36.7) | 101 (35.1)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Home Oxygen Therapy
Description: Duration of home oxygen use from time of randomization (baseline visit) to successful discontinuation of home oxygen therapy (HOT).
Time Frame: NICU discharge date until successful discontinuation of home oxygen therapy (HOT), up to 26 months.
Population: A total of 166 infants were weaned successfully from HOT using one of our two methods, and a total of 140 subjects completed all study procedures through six months of follow-up post discontinuation of HOT. A total of 30 subjects were not weaned using either method due to being lost to follow-up, withdrawing, or parents self-weaning subject.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Arm A:Standard Therapy | Arm B:RHO
Number analyzed (Participants) | 87 | 79
Days | 66 [42 to 113] | 58 [24 to 127]
Statistical Analysis 1: Comparison: Arm A:Standard Therapy vs Arm B:RHO; The trial was designed to have 97% power at a type I error rate of 5% to detect a 25% intervention effect with respect to the primary outcome. this was done using an independent sample t-test. P-value was calculated, and a p-value of 0.05 or less was interpreted as statistically significant result; Test type: Superiority; p < 0.03, t-test, 2 sided — A two-sided P-value of 0.05 or less was interpreted as a statistically significant result

2. Primary Outcome: Caregiver Quality of Life
Description: We will compare the difference between survey-derived quality-of-life scores, comparing parent response averages while on home oxygen therapy (HOT) versus 3 months post oxygen discontinuation scores in both arms. The infant scale is composed of 36 items comprising 5 dimensions. The item scaling is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores range from 0 to 100, with a higher score indicating a higher parent satisfaction and quality of life.
Time Frame: Monthly while on home oxygen therapy and at 3 months post discontinuation of therapy
Population: The final cohort included 196 infants, of those infants 105 parents completed at least one pre-parent satisfactory survey and one post-survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A:Standard Therapy | Arm B:RHO
Number analyzed (Participants) | 51 | 54
score on a scale
  Pre-Wean from HOT | 74.5 (16.3) | 70.4 (15.0)
  Post-Wean from HOT | 78.6 (18.6) | 75.9 (17.4)
Statistical Analysis 1: Comparison: Arm A:Standard Therapy vs Arm B:RHO; Power calculations were based on the primary analysis (t-test comparing changes). A sample size of 130 would have given 80% power, with 0.05 two sided type 1 error rate, to detect a 20% absolute difference in emotional role limitation on the PedsQL v2.0, which we considered to be statistically significant; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Participants With Respiratory-related Emergency Department Visits and Rehospitalizations
Description: We will assess rates of rehospitalization or ED visit throughout the weaning process and continue to assess until 6 months post discontinuation.
Time Frame: WIthin 6 months of discontinuation of home oxygen
Measure: Number; unit: participants
Arm/Group | Arm A:Standard Therapy | Arm B:RHO
Number analyzed (Participants) | 99 | 97
participants
  All Events | 41 | 25
  Serious Adverse Event | 28 | 19
  Life Threatening, ICU admission or Intubation (G4) | 7 | 6
  Hospitalization (G3) | 30 | 19
  Intervention without hospitalization | 39 | 26
  Event During Respiratory Virus Season | 29 | 17
  Event During Non-Respiratory Season | 26 | 15
  Respiratory Related Events | 26 | 20
  Non-Respiratory Related Events | 25 | 14

4. Secondary Outcome: Growth Parameters
Description: Growth measurements were taken at each monthly clinic visit while on oxygen. The average for weight z-score change was calculated for each subject while on oxygen therapy. After oxygen discontinuation, growth measurements were taken at the 1 month and 6 month post wean visits. These two measurements were again averaged for each patient. The weight z-score change was found in both arms for pre and post weaning from home oxygen therapy. The weight z-score indicates the number of standard deviations away from the mean a participants weight is. A z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Enrollment to 6 months post home oxygen therapy discontinuation
Population: We had data for 87 and 72 infants in the standard of care arm and RHO arm, respectively, during the O2 weaning process, and 80 and 73 infants after O2 discontinuation.
Measure: Mean (Standard Deviation); unit: Weight z-score change
Groups:
- Arm A: Standard of Care, Pre-Weaning; Arm B: Intervention Arm; Pre-Weaning: Growth assessments were documented at each monthly clinic visit while on oxygen. Infants who had at least one assessment were included in the analysis.
- Arm A: Standard of Care; Post-Weaning; Arm B: Intervention Arm; Post-Weaning: Growth assessments were documented at the one and six month follow-up visits. Infants who had at least one assessment were included in the analysis.
Arm/Group | Arm A: Standard of Care, Pre-Weaning | Arm B: Intervention Arm; Pre-Weaning | Arm A: Standard of Care; Post-Weaning | Arm B: Intervention Arm; Post-Weaning
Number analyzed (Participants) | 87 | 72 | 80 | 73
Weight z-score change | -0.13 (0.03) | -0.01 (0.03) | 0.02 (0.03) | 0.03 (0.03)

5. Secondary Outcome: Growth Parameters, Weight-for-length Z-score Change
Description: Growth measurements were taken at each monthly clinic visit while on oxygen. The average for weight for length z-score change was calculated for each subject while on oxygen therapy. After oxygen discontinuation, growth measurements were taken at the 1 month and 6 month post wean visits. These two measurements were again averaged for each patient. The weight for length z-score change was found in both arms for pre and post weaning from home oxygen therapy.The weight-for-length z-score indicates the number of standard deviations away from the mean a participants weight is. A z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Enrollment through 6 months post discontinuation of home oxygen therapy
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Weight-for-Length z-score change
Groups:
- Arm A: Standard of Care; Post-Weaning; Arm B: Intervention Arm; Post-Weaning: Growth assessments were documented at the one month and six month post wean follow-up visits. Infants who had at least one assessment in the follow-up period were included in the analysis.
Arm/Group | Arm A: Standard of Care, Pre-Weaning | Arm B: Intervention Arm; Pre-Weaning | Arm A: Standard of Care; Post-Weaning | Arm B: Intervention Arm; Post-Weaning
Number analyzed (Participants) | 87 | 72 | 80 | 73
Weight-for-Length z-score change | -0.17 (0.06) | -0.06 (0.07) | -0.14 (0.07) | 0.01 (0.07)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from enrollment until 6 months post home oxygen therapy discontinuation.
Description: Grade 1: No Intervention Grade 2: Intervention without hospitalization concomitant-drug/non-drug therapy Grade 3: Hospitalization (Serious Adverse Event) Grade 4: Life Threatening, ICU Admission, Intubation (Serious Adverse Event) Grade 5: Death (Serious Adverse Event)
Arm/Group | Arm A:Standard Therapy | Arm B:RHO
All-Cause Mortality (participants affected / at risk) | 41/99 | 26/97
Serious Adverse Events (participants affected / at risk) | 28/99 | 19/97
Other Adverse Events (participants affected / at risk) | 13/99 | 10/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A:Standard Therapy (N=99) | Arm B:RHO (N=97)
Viral Respiratory Event (Respiratory, thoracic and mediastinal disorders) | 16 (22) | 18 (20) — Former preterm infants are at an increased risk for respiratory adverse events and morbidity.
Feeding Issue/G-Tube Complication (Gastrointestinal disorders) | 8 (8) | 1 (2)
Other (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 0 (0) — Other serious adverse events related to prematurity
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A:Standard Therapy (N=99) | Arm B:RHO (N=97)
Respiratory Related Event (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT01994954/Prot_SAP_000.pdf